CLINICAL TRIAL: NCT06248944
Title: AIOCC Italian Registry on Head and Neck Carcinomas
Status: Recruiting | Type: Observational
Sponsor: Italian Head&Neck Society (Other)
Responsible Party: Sponsor
Other Study IDs: AIR Study
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational-retrospective and prospective — observational-retrospective and prospective

SUMMARY:
Multicentre, retrospective and prospective observational study aimed to set-up a clinical Italian registry in order to collect information on carcinoma of the Head and Neck.

DETAILED DESCRIPTION:
The registry plans to collect data on all patients treated or followed for Head and Neck cancer by the HCP of selected investigational sites in Italy.

Data will be entered manually by HCP staff of each investigational site in the study e-CRF in order to populate the AIR study database. Authorized HCPs will be provided with personal UserID and Password for the access to study eCRF.

For Data analysis an open-source system called Vantage6 will be used. It is a privacy preserving federated learning infrastructure for the secure exchange and analysis of incorporating data located at different sources. Queries will be issued to interrogate the database in order to have descriptive statistics and relevant information to plan the statistical analyses envisioned by the study protocol.

The registry data will support observational studies based on the second hand use of available data. Data collected for the AIR Study could be used also for global collaborative studies performed in Europe and outside the Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years old) diagnosed with carcinoma of the Head and Neck. The diagnosis should be done or verified by the expert site entering the information about the patient in the registry. Patients diagnosed with sarcomas and lymphomas are excluded.
2. Patients entering the HCP at any clinical phase of the disease (diagnosis, treatment of primary cancer, treatment of recurrence, treatment of M+ etc.). The HCP will collect information on the entire disease regardless of when it started to manage the patient. The HCP can choose, based on its resources, for how many patients will be able to collect the data.
3. New patients managed by the HCP from 2021 onwards + patients managed by the HCP, in active follow-up at the hospital

Exclusion Criteria:

1. Patients whose medical records are unavailable for review

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated or followed for Head and Neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
types of diagnostic and treatment patterns | From the enrollment to the end of the study (5 years)
  To document types of diagnostic and treatment patterns by all stages of disease and frequency, and proportion with which they are used in the different stages of Head and Neck cancer.

SECONDARY OUTCOMES:
proportion of patients in the different stage of disease | From the enrollment to the end of the study (5 years)
  To estimate the proportion of patients in the different stage of disease (TNM staging system 8^ edition) in the overall Head and Neck cancer patient population.
treatment outcomes | From the enrollment to the end of the study (5 years)
  To assess treatment outcomes in all patients by stage of disease
patients and disease characteristics | From the enrollment to the end of the study (5 years)
  To describe patients and disease characteristics (considering possibility of familiar occurrence).
benchmark values | From the enrollment to the end of the study (5 years)
  To find benchmark values for selected indicators (i.e., number of retrieved nodes, surgical complication, etc.) for surgical treatment
healthcare resource | From the enrollment to the end of the study (5 years)
  To evaluate healthcare resource utilization in the total population
prognostic factors | From the enrollment to the end of the study (5 years)
  To identify independent significant host-related prognostic factors and establish a more detailed prognostic classification for the growing population of Head and Neck cancer patients
between differences in mortality and differences in medical practice | From the enrollment to the end of the study (5 years)
  To prove the relationship between differences in mortality and differences in medical practice or medical organizations (subspecialty of the surgeon; type of hospital; management in the cancer network; conformity with clinical practice guidelines)
potential benefit | From the enrollment to the end of the study (5 years)
  To investigate the potential benefit for survival by classifying the detection of metastasis as early or late discoveries and by calculation of overall survival probabilities for both categories
immunization | From the enrollment to the end of the study (5 years)
  To determine the influence of immunization with vaccines preceding the removal of the primary tumor on prognosis of Head and Neck cancer patients, adjusting for stage, primary site, age, sex, particular treatment methods or patterns of referral
econometric approach | From the enrollment to the end of the study (5 years)
  To assess the links between costs and health outcomes using an econometric approach, taking into account confounding factors (stage, performance status, comorbidities, etc.).

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo
  - A.O.U. Careggi, Florence
  - P.O. 'Vito Fazzi', Lecce
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Fondazione CNAO, Pavia
  - Fondazione Policlinico Universitario 'Agostino Gemelli' IRCCS, Roma
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona

IPD SHARING:
Plan to Share IPD: No